CLINICAL TRIAL: NCT05599178
Title: Doppler Findings in the Fetal Cerebral Blood Vessels (VA/MCA) Within 24 Hours Before Delivery and Relation With Perinatal Outcome.
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66995
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Ultrasonography, Doppler; Obstetric Labor Complications
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Term gestation
  Interventions: Other: Ultrasound examination in early labor

INTERVENTIONS:
Other: Ultrasound examination in early labor — Combined trans-abdominal and trans-perineal ultrasound examination

SUMMARY:
1. Assess differences in flow patterns in the fetal cerebral blood vessels within 24 hours before delivery between fetuses with a normal vs. adverse perinatal outcome.
2. Explore maternal and/or fetal characteristics that might influence technical feasibility of doppler sonography of the fetal cerebral blood vessels in early labor at term.
3. Assess reliability of the technique by measuring intra- and inter-observer variation in a subset of participants.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Term gestation (37-42 weeks).
* Fetus in cephalic presentation.
* No known fetal chromosomal or (severe) congenital anomaly.
* Normally grown fetus (ultrasound scan demonstrating normal fetal growth between 30-37 weeks of gestation, defined as an estimated fetal weight/abdominal circumference > 10th centile or crossing <2 quartiles compared to earlier growth ultrasound).
* Absence of pre-existing doppler or amniotic fluid abnormalities.
* Normal fetal heart rate tracing / CTG (excluding pre-existing hypoxia).
* Admission in early spontaneous labor or induction of labor with expected delivery < 24 hours.
* Maternal age >= 18 years
* Willing to give written informed consent.

Exclusion Criteria:

* Advanced labor (> 4cm of cervical dilatation) at the time of admission on the labor ward.
* Severe pre-existing chronic maternal medical condition or poor obstetric history/antenatal complications associated with increased risk of adverse perinatal outcome (non-exhaustive e.g.: uncontrolled chronic hypertension, severe pre-eclampsia, uncontrolled (gestational) diabetes, maternal sepsis, major antepartum haemorrhage, intra-uterine infection, prolonged rupture of membranes > 18 hours, etc.).
* Intra-uterine fetal demise / death.
* Prelabour rupture of membranes with meconium-stained amniotic fluid.
* Patients not fulfilling all the inclusion criteria or refusing to give written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: "Low-risk" pregnant women
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in VPR (Vertebro-Placental Ratio) between fetuses/neonates with a composite perinatal outcome score < 3 / => 3 | VPR measured in early labor (=< 4cm of cervical dilatation) - perinatal outcome score assessed at delivery - timespan between both observations variable, expected <12 hours.

SECONDARY OUTCOMES:
Differences in other doppler parameters (PI VA, PI MCA, CPR) between fetuses/neonates with a composite perinatal outcome score < 3 / => 3. | VPR measured in early labor (=< 4cm of cervical dilatation) - perinatal outcome score assessed at delivery - timespan between both observations variable, expected <12 hours.
Differences in maternal and fetal characteristics between successful and unsuccessful doppler examinations (observations) of the fetal VA and MCA respectively. | Assessed in early labor (=< 4cm of cervical dilatation)

CONTACTS AND LOCATIONS:
Overall Officials: Jute Richter, MD, PhD, Principal Investigator — UZ Leuven / KU Leuven
Locations (1):
- University Hospitals Leuven, department of obstetrics and gynaecology, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided